CLINICAL TRIAL: NCT04450472
Title: Nonthyroidal Illness Syndrome in Patients With Short Bowel Syndrome
Brief Title: Nonthyroidal Illness Syndrome in SBS
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Wang Xinying, Director of the clinical nutrition center, Jinling Hospital, China
Other Study IDs: JinlingHospital
Record Dates: First submitted 2020-06-25; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Nonthyroidal Illness Syndrome; Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nonthyroidal illness syndrome (NTIS) is prevalent in critical illness; it is associated with poor outcomes. However, few studies have focused on the relationship between NTIS and short bowel syndrome (SBS). The aim of this study was to investigate the incidence, etiology, and prognosis of NTIS and its correlation in clinical variables in adult patients with SBS.

DETAILED DESCRIPTION:
Nonthyroidal illness syndrome (NTIS), also known as euthyroid sick syndrome or low triiodothyronine (T3) syndrome, is a condition characterized by decreased serum concentrations of T3 and low or normal plasma concentrations of thyroxine (T4) without a compensatory increase in the serum levels of thyroid stimulating hormone (TSH). However, such typical changes differ from those in primary or secondary thyroid disorders. NTIS refers to distortions in thyroid function without thyroid disease caused by various critical illnesses. This condition has been described in different acute and chronic disease states over the past 30 years, including sepsis, starvation, trauma, burns, myocardial infarction, Crohn's disease, enterocutaneous fistulas, chronic kidney disease, and major surgery.

Short bowel syndrome (SBS), the most common form of intestinal failure, is a rare condition resulting from the loss of portions of the intestine, typically because of extensive surgical resection or loss of intestinal function. Patients with SBS often stuffer from intestinal insufficiency or intestinal failure because they are unable to maintain fluid and nutrient balances on a normal diet. Therefore, SBS can cause various metabolic and physiologic disturbances, many of which are associated with growth, intestinal adaptation, and hormone secretion. Many previous studies of SBS have evaluated growth hormone, glucagon-like peptide-1, glucagon-like peptide-2, vitamin D and parathyroid hormone, peptide YY, and ghrelin. However, few studies have reported the association between SBS and the hypothalamic-pituitary-thyroid axis and its balance.

The present study was performed to evaluate the association of thyroid hormone disturbance and SBS in adult patients. Because NTIS is the main type of thyroid hormone disturbance, we further investigated the incidence, underlying mechanisms, and correlation with clinical variables and prognosis of NTIS in adult patients with SBS.

ELIGIBILITY:
Inclusion Criteria:

(1) Adult patients with SBS, defined as intestinal malabsorption disorder resulting from extensive bowel resection with a remnant small intestine length of greater than 200 cm, admitted to a clinical nutrition center.

-

Exclusion Criteria:

1. age less than 18 years;
2. previous history of thyroidal, hypophyseal or hypothalamic disease;
3. lactational or gestational period;
4. medication history of thyroidal hormone or antithyroid drugs;
5. craniocerebral injury;
6. attack of coronary heart disease, myocardial, or cerebral infarction in the past month;
7. intracranial infection or hemorrhage in the past month. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with SBS admitted to a clinical nutrition center in a tertiary referral hospital were identified to evaluate the incidence of NTIS and to explore its correlation with clinical variables and prognosis in adult patients.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-12-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Thyroid function index | Within one week of patients enrollment.
  Thyroid function assessment includes level of free triiodothyronine (FT3), total triiodothyronine (TT3), free thyroxin (FT4), total thyroxin (TT4), thyroid stimulating hormone (TSH).